CLINICAL TRIAL: NCT02677558
Title: The Impact of Obesity on Cardiac Function in Pregnancy
Acronym: CFOP
Status: Completed | Type: Observational
Sponsor: University of Cape Town (Other)
Responsible Party: Principal Investigator, Robert Dyer, Professor, University of Cape Town
Other Study IDs: 021/2016
Record Dates: First submitted 2016-02-04; First posted 2016-02-09 (Estimated); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Pregnancy; Obesity
Keywords: Pregnancy; Obesity; Echocardiography
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- CFOP obese: Transthoracic Echocardiography in pregnant women with a gestational age of greater or equal 36 weeks who have a BMI of greater or equal 40kg/m2 at the time point of inclusion into the study.
  Exclusion criteria: cardiac disease, on any cardiovascular drugs, pre-eclampsia or eclampsia.
  Interventions: Other: Transthoracic Echocardiography
- CFOP control: Transthoracic Echocardiography pregnant women with a gestational age of greater or equal 36 weeks who have a BMI of less or equal 30kg/m2 at the time point of inclusion into the study.
  Exclusion criteria: cardiac disease, on any cardiovascular drugs, pre-eclampsia or eclampsia
  Interventions: Other: Transthoracic Echocardiography

INTERVENTIONS:
Other: Transthoracic Echocardiography — Obese term pregnant women and term pregnant women of normal weight are both undergoing transthoracic echocardiography assessment to establish differences in cardiac function in pregnancy caused by obesity.

SUMMARY:
The purpose of this study is to determine the impact of obesity in pregnancy on maternal cardiac function. For this, morbidly obese term pregnant women (study group) and term pregnant women of normal weight are assessed by transthoracic echocardiography.

DETAILED DESCRIPTION:
INTRODUCTION:

The prevalence of obesity is increasing to alarming rates worldwide. The impact of obesity on cardiovascular health is well documented, but much less is known about the impact of obesity in pregnancy on maternal cardiac function. The aim of the current study is to investigate how the cardiovascular system of morbidly obese women adapts to the circulatory changes associated with pregnancy.

BACKGROUND:

Overweight and obesity is a major threat to global health. In 2013, 36.9% of all men and 38% of all women worldwide were overweight or obese as defined by a BMI of ≥25 kg/m2 or of ≥30 kg/m2 respectively. According to a systematic analysis for the Global Burden of Disease Study 2013, South Africa ranks third in a list of the world's most obese nations behind the United States and Mexico. The prevalence of overweight (BMI ≥25kg/m2) and obesity (BMI ≥30kg/m2) combined in the age group above 20 years is estimated to be 38.8% for men and 69.3% for women in South Africa. In the age group below 20 years, it is 18.8% for boys and 26.3% for girls. 42% of women above the age of 20 years and 9.6% of girls below 20 years are considered obese.

The impact of obesity on the structure and the function of the heart is well documented. Obesity is strongly associated with risk factors for the development of atherosclerotic disease such as hypertension, hyperlipidaemia, and diabetes. In addition, there is evidence that obesity in itself can lead to structural and functional changes in the heart. The following changes are commonly encountered in obesity:

1. Left ventricular remodelling: Many studies report that obesity is associated with an increase in left ventricular mass (LV mass). LV mass is commonly indexed against the body surface area (BSA). In the setting of significant obesity, LV mass/BSA is often normal or reduced, because the BSA increases more than the LV mass. Many investigators therefore choose to index LV mass to lean body mass, height or height raised to the power of 2.76. Recent studies agree that both wall thickness and cavity size seem to be increased in obesity, but wall thickness is increased to a greater extent, leading to a concentric pattern of left ventricular hypertrophy in obesity.
2. Right ventricular size: Only few studies have looked at the changes in the right ventricle in obesity. Wong et al. found mild increase in RV cavity size and wall thickness in uncomplicated obesity.
3. Left atrial size: Obesity is associated with an increase in left atrial size. Hypertension, volume overload and diastolic filling abnormalities commonly lead to an increase in left atrial size. All are commonly present in obesity.
4. Left ventricular systolic function: Recent studies report that LV ejection fraction is preserved in obesity or even above normal. There are, however subclinical contractile abnormalities which can already be found in obese children and adolescents comparable to those found in adult obese subjects.
5. Left ventricular diastolic function: The most common finding is that isovolumetric relaxation time is prolonged in obesity. Reduced tissue doppler velocities have also been reported.
6. Right ventricular function: Reduced RV systolic and diastolic function have been reported in individuals with a BMI ≥35kg/m2.

It is well established that obesity in pregnancy is a associated with an increased risk for thromboembolism, preeclampsia, postpartum haemorrhage, caesarean section and instrumental delivery. The impact of obesity during pregnancy might however reach even further. A well conducted retrospective study published in Hypertension this year found an association between obesity in pregnancy and premature mortality and morbidity from major cardiovascular events later in life. It is thought that the cardio-metabolic changes of obese pregnancy potentially unmask the patients at risk for cardiovascular events later in life.

Transthoracic echocardiography can detect subclinical alterations in cardiac structure and function. It is non-invasive and does not bear any risk for the mother or the baby. A routine assessment of the haemodynamic status in all obese pregnant women therefore has the potential to establish which women are at increased risk for haemodynamic complications during pregnancy and/or later in life. However, there have been only a limited number of studies on the haemodynamic changes in morbidly obese parturients as assessed by transthoracic echocardiography.

STUDY OBJECTIVES:

Hypothesis:

1. We hypothesise that cardiac dysfunction as determined by transthoracic echocardiography occurs more frequently in morbidly obese pregnant women than in pregnant women with normal BMI.
2. We hypothesise that the severity of the observed cardiac dysfunction correlates with the degree of obesity.

Aims:

1. To quantify the incidence of systolic and diastolic dysfunction and cardiac structural abnormalities in obese pregnant women at term.
2. To quantify the incidence of systolic and diastolic dysfunction and cardiac structural abnormalities in healthy term pregnant women with a normal BMI.
3. To quantify the severity of cardiac dysfunction and remodelling in obese pregnant women at term.

METHODOLOGY

Study design:

This prospective case control study will be carried out at Groote Schuur Maternity Clinic and Mowbray Maternity Hospital in Cape Town, South Africa.

Characteristics of study population:

We are aiming to recruit 40 obese pregnant, non-labouring women at term who fulfil the inclusion criteria. As controls, 40 healthy non-obese non-labouring term pregnant women will be recruited. Controls will be matched for age and ethnicity.

Recruitment:

Patients for the study group and the control group will be recruited from the antenatal clinic and antenatal wards.

Informed Consent:

Written informed consent will be obtained from all participants. Forms will be available in English and explained to the participants. The interview will be conducted in the participant's language of choice and a translator will assist with interpretation if required.

Data collection:

After enrolment in the study and informed consent, study patients and controls will undergo an echocardiographic examination as described below.

Demographic Data:

At the time point of enrolment, the following data will be recorded for all participants according to standard care in pregnancy:

* age
* gestational age and parity
* ethnicity
* height and weight
* blood pressure

Echocardiographic assessment:

A full standard echocardiographic assessment according to the protocol of the British Society of Echocardiography14 will be performed by an experienced investigator (passed European Echocardiography Examination), except subcostal views which are technically not feasible in pregnant women. In addition, a detailed right heart examination will be performed.

The examination will take place in the left lateral position to improve image quality and prevent obstruction of the inferior vena cava. A GE echocardiography machine will be used. For each acquisition, 3 cardiac cycles will be stored and analysed offline (after the examination) with Centricity Electronic Medical Records software developed by GE at a workstation at the Department of Anaesthesia/Cardiology. All echocardiographic assessments and offline analysis will be performed by one experienced investigators without blinding. Thereafter a second experienced investigator will review the images independently offline.

Schedule:

Data collection is planned to take place over a duration of 3 months in 2016.

Risks and Benefits:

Transthoracic echocardiography is a non-invasive procedure and safe for both the mother and the baby. No risk will arise due to participation in the study. The timing of the study will not interfere with routine clinical care.

If a cardiac condition is noted during the examination or any of the echocardiographic findings require a change to the planned care, this will be communicated to the patient's medical team without delay.

Participation in the study will therefore bring an additional clinical benefit to the mother at no additional risk.

Data handling and Confidentiality:

All demographic data pertaining to a participant will be collected on a standardised form.

Each participant will be assigned a unique study number. The echocardiography data will be stored on the GE echocardiography machine using this number only, with no identifying information. From here the data will be exported to the hospital based echocardiography data system for analysis (Centricity Electronic Medical Records). The participants are thus de-linked from their hospital admission numbers and confidentiality is protected. The records can only be accessed with an assigned login from Groote Schuur hospital that will only be available to the approved users of the Centricity system.

A record of hospital admission numbers will be maintained to correlate echocardiography data with clinical data and allow the patient's medical team to be informed of any relevant pathology that may impact patient care. The Principal Investigator will have access to the record log and this information will not be made available outside the University of Cape Town.

Study records that identify a patient are kept confidential as required by law. Privacy regulations provide safeguards for privacy, security and authorised access. Except when required by law, no data will identify the patient in the study records. The data collected remains the intellectual property of the University of Cape Town.

Data Analysis:

Demographic and obstetrics data will be displayed as mean and standard deviation, median with interquartile ranges, or number and percentage as appropriate. Analysis of recorded transthoracic echocardiography variables and heart rate and blood pressure will be made using analysis of variance (ANOVA) and a General Linear Model with significant p value defined as < 0.05 after performing F tests on the collected data. Pearson's correlation will be used to assess the strength of the linear relationship between variables. The null hypothesis will be rejected if critical p < 0.05 for each of the variables.

ELIGIBILITY:
Inclusion Criteria:

* BMI >/= 35kg/m2 for study group and </= 30kg/m2 for control group
* uncomplicated singleton term pregnancy

Exclusion Criteria:

* any comorbidities affecting cardiac function
* receiving any cardiovascular drugs
* in active labour
* inability to give informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Healthy obese pregnant, non-labouring women at term who fulfil the inclusion criteria will be recruited into the study group. As controls, healthy non-obese non-labouring term pregnant women will be recruited. Controls will be matched for age and ethnicity.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2016-01; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Incidence of systolic and diastolic cardiac dysfunction in morbidly obese pregnant women compared to term pregnant women of normal weight through transthoracic echocardiography. | At inclusion into study

SECONDARY OUTCOMES:
Correlation of degree of cardiac dysfunction in morbidly obese term pregnant women with BMI | At inclusion into study

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Dyer, Medicine, Principal Investigator — University of Cape Town
Locations (1):
- University of Cape Town; Groote Schuur Hospital, Cape Town, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abel ED, Litwin SE, Sweeney G. Cardiac remodeling in obesity. Physiol Rev. 2008 Apr;88(2):389-419. doi: 10.1152/physrev.00017.2007. PMID 18391168
- [Background] Wong CY, O'Moore-Sullivan T, Leano R, Hukins C, Jenkins C, Marwick TH. Association of subclinical right ventricular dysfunction with obesity. J Am Coll Cardiol. 2006 Feb 7;47(3):611-6. doi: 10.1016/j.jacc.2005.11.015. Epub 2006 Jan 18. PMID 16458145
- [Background] Powell BD, Redfield MM, Bybee KA, Freeman WK, Rihal CS. Association of obesity with left ventricular remodeling and diastolic dysfunction in patients without coronary artery disease. Am J Cardiol. 2006 Jul 1;98(1):116-20. doi: 10.1016/j.amjcard.2006.01.063. Epub 2006 May 6. PMID 16784933
- [Background] Peterson LR, Waggoner AD, Schechtman KB, Meyer T, Gropler RJ, Barzilai B, Davila-Roman VG. Alterations in left ventricular structure and function in young healthy obese women: assessment by echocardiography and tissue Doppler imaging. J Am Coll Cardiol. 2004 Apr 21;43(8):1399-404. doi: 10.1016/j.jacc.2003.10.062. PMID 15093874
- [Background] de Simone G, Kizer JR, Chinali M, Roman MJ, Bella JN, Best LG, Lee ET, Devereux RB; Strong Heart Study Investigators. Normalization for body size and population-attributable risk of left ventricular hypertrophy: the Strong Heart Study. Am J Hypertens. 2005 Feb;18(2 Pt 1):191-6. doi: 10.1016/j.amjhyper.2004.08.032. PMID 15752946
- [Background] de Simone G, Devereux RB, Roman MJ, Alderman MH, Laragh JH. Relation of obesity and gender to left ventricular hypertrophy in normotensive and hypertensive adults. Hypertension. 1994 May;23(5):600-6. doi: 10.1161/01.hyp.23.5.600. PMID 8175168
- [Background] Wong CY, O'Moore-Sullivan T, Leano R, Byrne N, Beller E, Marwick TH. Alterations of left ventricular myocardial characteristics associated with obesity. Circulation. 2004 Nov 9;110(19):3081-7. doi: 10.1161/01.CIR.0000147184.13872.0F. Epub 2004 Nov 1. PMID 15520317
- [Background] Reidy J, Russell R. CMACE 2006-2008. Int J Obstet Anesth. 2011 Jul;20(3):208-12. doi: 10.1016/j.ijoa.2011.04.004. No abstract available. PMID 21641202
- [Background] Lee KK, Raja EA, Lee AJ, Bhattacharya S, Bhattacharya S, Norman JE, Reynolds RM. Maternal Obesity During Pregnancy Associates With Premature Mortality and Major Cardiovascular Events in Later Life. Hypertension. 2015 Nov;66(5):938-44. doi: 10.1161/HYPERTENSIONAHA.115.05920. Epub 2015 Sep 14. PMID 26370890
- [Background] Dennis AT, Castro JM, Ong M, Carr C. Haemodynamics in obese pregnant women. Int J Obstet Anesth. 2012 Apr;21(2):129-34. doi: 10.1016/j.ijoa.2011.11.007. Epub 2012 Feb 11. PMID 22326199
- [Background] Ng M, Fleming T, Robinson M, Thomson B, Graetz N, Margono C, Mullany EC, Biryukov S, Abbafati C, Abera SF, Abraham JP, Abu-Rmeileh NM, Achoki T, AlBuhairan FS, Alemu ZA, Alfonso R, Ali MK, Ali R, Guzman NA, Ammar W, Anwari P, Banerjee A, Barquera S, Basu S, Bennett DA, Bhutta Z, Blore J, Cabral N, Nonato IC, Chang JC, Chowdhury R, Courville KJ, Criqui MH, Cundiff DK, Dabhadkar KC, Dandona L, Davis A, Dayama A, Dharmaratne SD, Ding EL, Durrani AM, Esteghamati A, Farzadfar F, Fay DF, Feigin VL, Flaxman A, Forouzanfar MH, Goto A, Green MA, Gupta R, Hafezi-Nejad N, Hankey GJ, Harewood HC, Havmoeller R, Hay S, Hernandez L, Husseini A, Idrisov BT, Ikeda N, Islami F, Jahangir E, Jassal SK, Jee SH, Jeffreys M, Jonas JB, Kabagambe EK, Khalifa SE, Kengne AP, Khader YS, Khang YH, Kim D, Kimokoti RW, Kinge JM, Kokubo Y, Kosen S, Kwan G, Lai T, Leinsalu M, Li Y, Liang X, Liu S, Logroscino G, Lotufo PA, Lu Y, Ma J, Mainoo NK, Mensah GA, Merriman TR, Mokdad AH, Moschandreas J, Naghavi M, Naheed A, Nand D, Narayan KM, Nelson EL, Neuhouser ML, Nisar MI, Ohkubo T, Oti SO, Pedroza A, Prabhakaran D, Roy N, Sampson U, Seo H, Sepanlou SG, Shibuya K, Shiri R, Shiue I, Singh GM, Singh JA, Skirbekk V, Stapelberg NJ, Sturua L, Sykes BL, Tobias M, Tran BX, Trasande L, Toyoshima H, van de Vijver S, Vasankari TJ, Veerman JL, Velasquez-Melendez G, Vlassov VV, Vollset SE, Vos T, Wang C, Wang X, Weiderpass E, Werdecker A, Wright JL, Yang YC, Yatsuya H, Yoon J, Yoon SJ, Zhao Y, Zhou M, Zhu S, Lopez AD, Murray CJ, Gakidou E. Global, regional, and national prevalence of overweight and obesity in children and adults during 1980-2013: a systematic analysis for the Global Burden of Disease Study 2013. Lancet. 2014 Aug 30;384(9945):766-81. doi: 10.1016/S0140-6736(14)60460-8. Epub 2014 May 29. PMID 24880830
- See also: A Minimum Dataset for a Standard Transthoracic Echocardiogram from the British Society of Echocardiography Education Committee — http://www.google.ch/url?sa=t&rct=j&q=&esrc=s&source=web&cd=1&ved=0ahUKEwikyqGc_dbKAhWIVhQKHTcsCjoQFggjMAA&url=http%3A%2F%2Fwww.bsecho.org%2Ftte-minimum-dataset%2F&usg=AFQjCNG_CvnmSvI89u4TPSiKXawoxpoMog&bvm=bv.113034660,d.ZWU